CLINICAL TRIAL: NCT03060551
Title: Safety, Tolerability and Potential Efficacy of Injection of Autologous Adipose-derived Stromal Vascular Fraction in the Finger of Systemic Sclerosis Patients
Brief Title: Injection of Autologous Adipose-derived Stromal Vascular Fraction in the Finger of Systemic Sclerosis Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Suk-Ho Moon (Other)
Responsible Party: Sponsor-Investigator, Suk-Ho Moon, Assistant Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SVF treatment in SSc
Record Dates: First submitted 2016-11-09; First posted 2017-02-23 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Systemic Sclerosis
Keywords: stromal vascular fraction; hand disability; mesenchymal stem cells; phase I trial
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Intervention Model Description: Systemic sclerosis patients with hand disability, planning 24 weeks of follow-up period Autologous adipose tissue-derived stromal vascular fraction(SVF) injected into the subcutaneous tissue of each finger in contact with neurovascular pedicles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SVF injection (Experimental): SVF was obtained from lipoaspirates, using an automated processing system, and subsequently injected into the subcutaneous tissue of each finger in contact with neurovascular pedicles
  Interventions: Procedure: SVF injection

INTERVENTIONS:
Procedure: SVF injection — SVF is increasingly recognised as an easily accessible source of regenerative cells with therapeutic potential in ischaemic or autoimmune disease. We aimed to measure for the first time the safety, tolerability and potential efficacy of autologous SVF cells local injections in patients with systemic sclerosis

SUMMARY:
This study outlines the safety of the autologous SVF cells injection in the hands of patients with SSc. Preliminary assessments at 6 months will suggest potential efficacy needing confirmation in a randomised placebo-controlled trial on a larger population

DETAILED DESCRIPTION:
In patients with systemic sclerosis(scleroderma, SSc), impaired hand function greatly contributes to disability and reduced quality of life, and is insufficiently relived by currently available therapies. Adipose tissue-derived stromal vascular fraction (SVF) is increasingly recognized as an easily accessible source of regenerative cells with therapeutic potential in ischaemic or autoimmune disease. The investigators aimed to measure for the first time the safety, tolerability, and potential efficacy of autologous SVF cells local injections in patients with SSc with hand disability.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 year old
* Cochin Hand Function Scale (CHFS) > 20/90

Exclusion Criteria:

* new vasodilators or immunosuppressive therapy for SSc in the 3 months prior to enrolment
* new vasodilators or immunosuppressive therapy for SSc during the 6-month follow-up
* clinical or radiological signs of digital infection
* positive status for HIV
* positive status for hepatitis B or C
* positive status for human T-cell leukemia virus 1-2
* positive status for syphilis
* pregnancy
* BMI less than 17kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suk-Ho Moon, MD, PhD, Study Director — Seoul St. Mary's Hospital; Seung-Ki Kwok, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, College of Medicine, The Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park Y, Lee YJ, Koh JH, Lee J, Min HK, Kim MY, Kim KJ, Lee SJ, Rhie JW, Kim WU, Park SH, Moon SH, Kwok SK. Clinical Efficacy and Safety of Injection of Stromal Vascular Fraction Derived from Autologous Adipose Tissues in Systemic Sclerosis Patients with Hand Disability: A Proof-Of-Concept Trial. J Clin Med. 2020 Sep 19;9(9):3023. doi: 10.3390/jcm9093023. PMID 32961802

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July 2018 and December 2019, a total of twenty subjects were enrolled in this single center, open label, phase I trial.
Pre-assignment Details: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection.
Groups:
- SVF Injection Group: Participants received SVF treatment, and were fully followed-up for the whole scheduled period for clinical assessment. SVF extraction and injection were performed in outpatient setting within at least 1 month after baseline evaluation. All patients were regulary assessed for intervention-related adverse events and clinical efficacies at 2 weeks (2W), 6 weeks (6W), 12 weeks (12W) and 24 weeks (24W) after their procedure.
Period: Overall Study
Arm/Group | SVF Injection Group
Started | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | SVF Injection
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  years
    number analyzed (Participants) | 18
    (all) | 47 [42 to 57]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    Female | 15
    Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 20
Body mass index (BMI) kg/m2 [Median (Inter-Quartile Range); unit: kg/m2] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  kg/m2
    number analyzed (Participants) | 18
    (all) | 21.5 [18.2 to 23.1]
Disease duration (years) [Median (Inter-Quartile Range); unit: years] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  years
    number analyzed (Participants) | 18
    (all) | 6 [1 to 17]
Reynaud's phenomenon duration [Median (Inter-Quartile Range); unit: years] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  years
    number analyzed (Participants) | 18
    (all) | 9 [4 to 17]
Smoking history (Current or ex-) [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 3
Interstitial lung disease [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 10
Types of cutaneous manisfetations (diffuse or limited) [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    Diffuse | 8
    Limited | 10
Hand dominance (right) [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 18
Pulmonary hypertension [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 1
History of renal crisis [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 1
Diabetes mellitus [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 0
Hypertension [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 0
Osteoporosis [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 6
Medication status (calcium channel blocker) [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 9
Medication status (prostacyclin) [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 2
Medication status (Aloprostadil) [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 3
Medication status (Endothelial receptor antagonist)) [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 1
Medication status (Azathioprine) [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 5
Medication status (Glucocorticoid) [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 13
Medication status (Methotrexate) [Count of Participants; unit: Participants] — Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 8
Anti-nuclear antibody [Count of Participants; unit: Participants] — Antinuclear autoantibodies are present in more than 90% of patients with systemic sclerosis (SSc). The presence of antinuclear antibodies is a central feature of systemic sclerosis. Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 18
Anti-centromere antibody [Count of Participants; unit: Participants] — Anti-centromere antibodies are autoantibodies specific to centromere function. They occur in some autoimmune diseases, freqently in limited systemic scleroderma. Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 4
Anti-Scl70 antibody [Count of Participants; unit: Participants] — Anti-Scl-70 autoantibodies are found in 20~35% of patients with systemic sclerosis, mainly in those with the diffuse form of the disease. Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 13
Anti-Ro/SSA antibody [Count of Participants; unit: Participants] — Anti-Ro/SSA antibodies are anti-nuclear autoantibodies that are associated with many autoimmune diseases. Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 4
Anti-U1 RNP antibody [Count of Participants; unit: Participants] — Anti-U1 RNP antibody is generally known to be a serological marker for mixed connective tissue disease, but can be detected also in patients with definite systemic sclerosis. Population: Among the initially enrolled patients, one patient refused further procedures after baseline evaluation, while another patient dropped out due to complications during local anesthesia right before SVF injection (one patient dropout due to dizziness after lidocaine injection where the prepared SVF was discarded).
  Participants
    number analyzed (Participants) | 18
    (all) | 5

OUTCOME MEASURES:

1. Primary Outcome: Raynaud's Condition Scale
Description: The severity of Raynaud's phenomenon was assessed using the Raynaud's condition scale (ranging 0 to 10, with higher scores representing more severe Raynaud's phenomenon)
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  baseline | 5 [1.8 to 7.3]
  2 weeks | 5 [2 to 7.3]
  6 weeks | 6.5 [4.5 to 7.0]
  12 weeks | 3 [2 to 5]
  24 weeks | 6 [2 to 7.5]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — Because most efficacy data consisted of non-parameteric variables, results were shown as median values and interquartile range. The Wilcoxon signed-rank test was performed to analyze differences between baseline and at 2W, 6W, 12W and 24W, respectively, using IBM-SPSS Statistics version 24.0 (SPSS Inc., Chicago, IL, USA). Statistical significance was considered at p < 0.05. Safety profiles were descriptively analyzed; p = 0.256, Wilcoxon (Mann-Whitney) — p value (24 weeks-baseline)

2. Primary Outcome: Hand Visual Analogue Scale
Description: Hand pain was assessed using the Hand visual analogue scale (ranging 0 to 10, with higher scores representing more severe pain)
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  baseline | 5 [2.5 to 5]
  2 weeks | 4 [2 to 5]
  6 weeks | 5 [3.5 to 6]
  12 weeks | 4 [2 to 6]
  24 weeks | 5 [2.5 to 7]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.682, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

3. Primary Outcome: Colchin Hand Function Scale
Description: The Colchin hand function scale (CHFS, ranging 0 to 90, with higher scores representing more deteriorated hand function) scores
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 7.5 [3.3 to 21.8]
  2 weeks | 14 [0 to 23.3]
  6 weeks | 16 [1.5 to 30.3]
  12 weeks | 18 [1 to 27.5]
  24 weeks | 17 [1.5 to 33]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.151, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

4. Primary Outcome: Kapandji Score (Ranging 0 to 10) - Dominant Hand
Description: Kapandji score (ranging 0 to 10) is validated measures in past studies as outcomes for hand disability. The Kapandji score is a tool useful for assessing the opposition of the thumb, based on where on their hand the patient is able to touch with the tip of their thumb. A score of 0 indicates no opposition, a score of 10 indicates maximal opposition.
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 9 [8 to 9]
  2 weeks | 9 [8 to 9]
  6 weeks | 9 [8 to 9]
  12 weeks | 9 [8 to 9]
  24 weeks | 8 [8 to 9]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.516, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

5. Primary Outcome: Kapandji Score (Non-dominant Hand)
Description: as for outcome 4
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 9 [8 to 9]
  2 weeks | 9 [8 to 9]
  6 weeks | 9 [8.8 to 9]
  12 weeks | 9 [8 to 9]
  24 weeks | 9 [8 to 9]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p > 0.999, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

6. Primary Outcome: Disease-related QOL (Quality of Life) : EuroQol-5 Dimensions Time Trade-off (EQ-5D TTO)
Description: Disease-related QOL (quality of life) was measured by EuroQol-5 dimensions time trade-off (EQ-5D TTO, ranging 0 to 1, with higher values representing better QOL) values
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 0.807 [0.709 to 0.880]
  2 weeks | 0.804 [0.723 to 0.858]
  6 weeks | 0.779 [0.685 to 0.888]
  12 weeks | 0.801 [0.715 to 0.862]
  24 weeks | 0.888 [0.710 to 0.930]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.034, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

7. Primary Outcome: Disease-related QOL (Quality of Life) : EuroQol Visual Analog Scale (EQ VAS)
Description: Disease-related QOL (quality of life) : EuroQol visual analog scale (EQ VAS, ranging 0 to 100, with higher scores representing better QOL)
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 70 [50 to 81]
  2 weeks | 68 [50 to 80]
  6 weeks | 70 [50 to 75]
  12 weeks | 80 [70 to 88]
  24 weeks | 80 [55 to 83]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.656, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

8. Primary Outcome: Disease-related QOL (Quality of Life) : Health Assessment Questionnaire (HAQ)
Description: Disease-related QOL (quality of life) : health assessment questionnaire (HAQ, ranging 0 to 3, with higher scores meaning lower QOL)
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 1.000 [0.219 to 1.406]
  2 weeks | 0.938 [0.219 to 1.375]
  6 weeks | 1.000 [0.000 to 1.563]
  12 weeks | 0.750 [0.063 to 1.438]
  24 weeks | 0.625 [0.188 to 1.313]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.096, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

9. Primary Outcome: The Degree of Hand Edema (Right)
Description: The finger circumferences of the second to the fifth fingers measured in the middle portion of each proximal phalanx were used to assess the degree of hand edema
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
cm
  Baseline | 5.9 [5.7 to 6.4]
  2 weeks | 5.9 [5.5 to 6.4]
  6 weeks | 6.0 [5.6 to 6.3]
  12 weeks | 6.0 [5.7 to 6.4]
  24 weeks | 5.9 [5.7 to 6.3]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.019, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

10. Primary Outcome: The Degree of Hand Edema (Left)
Description: as for outcome 9
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
cm
  Baseline | 5.9 [5.6 to 6.2]
  2 weeks | 5.8 [5.5 to 6.3]
  6 weeks | 5.8 [5.5 to 6.3]
  12 weeks | 5.9 [5.6 to 6.2]
  24 weeks | 5.9 [5.6 to 6.3]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.050, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

11. Secondary Outcome: Changes of Nailfold Capillary Microscopic Findings (Irregularly Enlarged Capillaries)
Description: In order to assess the severity of microangiopathies in both fingers, a semiquantitative scoring system for nailfold capillary microscopic findings was adopted. A total of six parameters (irregularly enlarged capillaries, giant capillaries, hemorrhages, loss of capillaries, disorganization of the vascular array and capillary ramifications) were measured using the semiquantitative manner on the scale ranging 0 to 3, indicating more severe as scores were higher. Each parameter was scored for four fingers of both hands, except thumbs, and the median score value of each parameter in both hands was finally presented.
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 0.938 [0.594 to 1.969]
  2 weeks | 1.313 [0.469 to 1.813]
  6 weeks | 1.000 [0.5000 to 1.813]
  12 weeks | 1.250 [0.750 to 1.625]
  24 weeks | 1.125 [0.688 to 1.563]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.372, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

12. Secondary Outcome: Changes of Nailfold Capillary Microscopic Findings (Giant Capillaries)
Description: as for outcome 11
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 0.125 [0.000 to 1.375]
  2 weeks | 0.000 [0.000 to 0.656]
  6 weeks | 0.063 [0.000 to 0.688]
  12 weeks | 0.000 [0.000 to 0.625]
  24 weeks | 0.125 [0.000 to 0.313]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.024, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

13. Secondary Outcome: Changes of Nailfold Capillary Microscopic Findings (Hemorrhages)
Description: as for outcome 11
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 0.000 [0.000 to 0.125]
  2 weeks | 0.000 [0.000 to 0.063]
  6 weeks | 0.000 [0.000 to 0.094]
  12 weeks | 0.000 [0.000 to 0.188]
  24 weeks | 0.125 [0.000 to 0.313]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.188, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

14. Secondary Outcome: Changes of Nailfold Capillary Microscopic Findings (Loss of Capillaries)
Description: as for outcome 11
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 2.188 [1.469 to 2.406]
  2 weeks | 2.063 [1.438 to 2.500]
  6 weeks | 2.063 [1.625 to 2.344]
  12 weeks | 2.000 [1.438 to 2.563]
  24 weeks | 2.250 [1.313 to 2.563]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.372, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

15. Secondary Outcome: Changes of Nailfold Capillary Microscopic Findings (Disorganization of the Vascular Array)
Description: as for outcome 11
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 0.688 [0.188 to 1.625]
  2 weeks | 0.688 [0.563 to 1.906]
  6 weeks | 0.688 [0.000 to 1.688]
  12 weeks | 0.875 [0.000 to 1.875]
  24 weeks | 0.375 [0.000 to 1.938]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.633, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

16. Secondary Outcome: Changes of Nailfold Capillary Microscopic Findings (Capillary Ramifications)
Description: as for outcome 11
Time Frame: Baseline, 2 weeks, 6 weeks, 12 weeks, 24 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SVF Injection Group
Number analyzed (Participants) | 18
score on a scale
  Baseline | 0.125 [0.000 to 0.375]
  2 weeks | 0.125 [0.000 to 0.438]
  6 weeks | 0.000 [0.000 to 1.688]
  12 weeks | 0.063 [0.000 to 0.594]
  24 weeks | 0.125 [0.000 to 0.375]
Statistical Analysis 1: Comparison: SVF Injection Group; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.380, Wilcoxon (Mann-Whitney) — p-value (24 weeks-baseline)

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Description: No serious adverse events occurred throughout study.
Groups:
- SVF Injection Group: Participants received SVF treatment. All patients were regulary assessed at 2 weeks (2W), 6 weeks (6W), 12 weeks (12W) and 24 weeks (24W) after their procedure.
Arm/Group | SVF Injection Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SVF Injection Group (N=20)
Transient paresthesia in liposuction lesions (Injury, poisoning and procedural complications) | 1 (1)
Dizziness after lidocaine injection (Injury, poisoning and procedural complications) | 1 (1)
Transient pallor in finger after injection (Injury, poisoning and procedural complications) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT03060551/Prot_SAP_000.pdf